CLINICAL TRIAL: NCT06989463
Title: Complementary Behavioral Interventions To Remediate Cognitive Impairment or Emotional Distress in Cancer Survivors: A Pilot Study
Brief Title: Complementary Behavioral Interventions To Remediate Cognitive Impairment or Emotional Distress in Cancer Survivors
Acronym: COPILOT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: COPILOT; NCI-2025-05387 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2025-05-08; First posted 2025-05-25 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Survivors of Childhood Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (EX) plus Cognitive Training (CT) (Active Comparator): Adult survivor of childhood cancer enrolled in St. Jude Life Cohort (SJLIFE) at least five years from diagnosis.
  Participants pre-identified as cognitively impaired will be assigned to the EX+CT arm
  Interventions: Other: 12 Week Exercise Intervention; Other: Cognitive Training Intervention
- Exercise (EX) plus Mindfulness Practice (MP) (Active Comparator): Adult survivor of childhood cancer enrolled in St. Jude Life Cohort (SJLIFE) at least five years from diagnosis.
  Participants pre-identified as emotionally impaired will be assigned to the EX+MP arm.
  Interventions: Other: 12 Week Exercise Intervention; Other: Mindfulness practice intervention

INTERVENTIONS:
Other: 12 Week Exercise Intervention — Participants will be provided with the results of their physical functioning and fitness assessments and will receive an individually tailored exercise prescription, written by an exercise specialist and approved by the study physician. The prescription will include aerobic and strengthening components designed to progress persons gradually to 150-300 minutes of the equivalent of moderate aerobic activity and twice weekly strengthening106 over 12 weeks.
Other: Cognitive Training Intervention — Participants will complete cognitive training with Lumosity (Lumos Labs, Inc.; San Francisco, California; cognitive training program). This computer-based training consists of games focused on specific executive function skills (shifting attention, working memory, verbal fluency, problem solving). Each 20-minute session includes five games focused specifically on these executive functioning skills.
  Participants will be prescribed three 20-minute sessions each week for 12-weeks.
  Arms: Exercise (EX) plus Cognitive Training (CT)
Other: Mindfulness practice intervention — The mindfulness practice intervention is a modified version of the University of California at Los Angeles Mindfulness Awareness Research Center's Mindful Awareness Practices designated to be remotely delivered.
  during odd weeks, participants will watch the educational lecture video once and practice meditation daily. During even weeks, they will review the educational video as needed and continue daily meditation practice.
  Arms: Exercise (EX) plus Mindfulness Practice (MP)

SUMMARY:
Childhood cancer survivors are at risk for accelerated aging due to the specific treatments they have received to cure their cancer. Several interventions, including exercise, cognitive training, and mindfulness practice, have been developed and studied for effectiveness among participants in the St. Jude Lifetime Cohort (SJLIFE) to mitigate these effects. The interventions offered thus far have not included two components at the same time.

The purpose of this study is to determine whether or not adult cancer survivors enrolled in SJLIFE will participate in two interventions at the same time. The combined interventions will include exercise plus cognitive training or exercise plus mindfulness practice. Each intervention will be conducted over a 12-week period. Participants will also be asked to complete follow-up testing after the 12-week intervention period is completed.

Primary Objectives

• To determine the acceptability of a two-component intervention (exercise (EX) plus cognitive training (CT) or exercise (EX) plus mindfulness practice (MP)) among survivors of childhood cancer with either cognitive impairment or emotional distress.

Hypotheses:

* 45% of those approached for participation in each arm of this study will enroll on the study.
* Among those who enroll, 70% will complete the follow-up testing at 12 weeks.
* Among those who completed the follow-up testing, the mean attendance to the intervention sessions will be 70% on each of their two interventions. That is, they will complete 70% of exercise sessions and 70% of either cognitive training or mindfulness practice.
* To identify barriers and facilitators to intervention adherence.

Hypotheses:

* Participants will identify features of the study processes that either facilitate or discourage adherence.
* Participants will identify features of the intervention technology and intervention components that either facilitate or discourage adherence.
* Participants will identify personal factors that facilitate or discourage adherence.

DETAILED DESCRIPTION:
The study will recruit survivors from the SJLIFE cohort who have completed a recent SJLIFE campus visit and were pre-identified as either cognitively (by self-report on Childhood Cancer Survivor Study (CCSS) NCQ) or emotionally impaired (by self-report on the BSI). We plan to recruit 10 survivors from each impairment group. All survivors will be at least five years from diagnosis.

Participants will be assigned to one of two interventions - 1) (exercise (EX) plus cognitive training (CT) or 2) exercise (EX) plus mindfulness practice (MP).

Those pre-identified as cognitively impaired will be assigned to the EX+CT arm and those pre-identified as emotionally impaired will be assigned to the EX+MP arm.

The make up in each of the two study interventions will include 3 survivors aged 18-29 years, 4 survivors aged 30-39 years, and 3 survivors aged 40 years or older. Additionally, each intervention will include 5 males and 5 females and at least 4 survivors that report either non-Hispanic black or Hispanic race/ethnicity.

Potentially eligible participants have already been screened for physical, cognitive, and emotional impairments based on data previously collected at a recent SJLIFE campus visit. All participants identified will engage in <150-minutes/week of moderate/vigorous physical activity and are either cognitively or emotionally impaired (as indicated on a recently completed neurocognitive or emotional health questionnaire).

Each arm will participate in a 12-week intervention period. All participants will receive the necessary equipment to complete the remote assessments (e.g., pregnancy test if female, laptop configured with access to exercise platform, cognitive training and mindfulness practice materials, pulse oximeter, blood pressure monitor, etc.) as well as exercise equipment (e.g., exercise mat, resistance bands). Each participant will complete a remote assessment before and after the intervention period.

All participants will receive an individually tailored exercise prescription, written by an exercise specialist and approved by the study physician. The prescription will include aerobic and strengthening components designed to progress the participants gradually to 150-300 minutes of the equivalent of moderate aerobic activity and twice weekly strengthening over 12 weeks.

Participants assigned to cognitive training will use a computer-based training which consists of games focused on specific executive function skills (shifting attention, working memory, verbal fluency, problem solving). Participants will be prescribed three 20-minute sessions each week for 12-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants enrolled in St. Jude Lifetime Cohort (SJLIFE) >18 years of age.
* Participant has been pre-identified as both physically impaired (T score ≤45 on the physical function and/or role physical subscales of the Medical Outcomes Survey Short Form 36 (SF-36)), and either cognitively (standard score >84th percentile on the Childhood Cancer Survivor Study Neurocognitive Questionnaire) or emotionally impaired (T scored score ≥ 63 on the Brief Symptom Inventory) from the most recently completed SJLIFE survey questionnaires.
* Participant self-reports participating in <150 minutes of moderate to vigorous physical activity per week (Centers for Disease Control Physical Activity Guidelines for Americans).
* Participant has been medically cleared to participate in physical activity.
* Participant verbalizing understanding of the directions to use the digital platform on provided laptop/tablet.

Exclusion Criteria:

* Participant cannot speak, read, and/or understand English.
* Participant is a woman and currently pregnant.
* Participant reports engaging in mindfulness-based training or continuously practiced mindfulness techniques over the past 6 weeks.
* Participant has an estimated intelligence score (FSIQ) <80.
* Participant has a diagnosis of post-traumatic stress disorder, major psychiatric condition, and/or history of suicidal ideation or self-harm.
* Participant reports alcohol or drug abuse in the past year (Alcohol Use Disorders Identification Test (AUDIT) >=13/women and >=15/men or Drug Abuse Screen Test (DAST) -10>3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate (%) | Through study completion or an average of 24 months
  The percentage of the number of participants approached for participation compared to those who enroll on study
Follow up completion rate (%) | Through study completion or an average of 24 months
  The percentage of the number of participants who complete the 12-week testing compared to who enroll on study
Intervention adherence rate for those participants who complete the final follow up visit (%) | Through study completion or an average of 24 months
  The percentage of the intervention sessions attended v offered (n=24)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten K Ness, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the ClinicalTrials.gov (CTG) website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: Description Clinical Trials Open at St. Jude — http://www.stjude.org/protocols